CLINICAL TRIAL: NCT06661759
Title: Clinic-based and Technology-Supported Sleep Intervention for Pediatric Epilepsy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 202402064RINE
Record Dates: First submitted 2024-10-24; First posted 2024-10-28 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2025-11

CONDITIONS: Epilepsy
MeSH Terms: conditions — Epilepsy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental intervention group (Experimental): standard pediatric neurology care plus a hybrid in-person and digital sleep education program
  Interventions: Behavioral: Clinic-based and technology-supported sleep intervention
- Usual care group (No Intervention): standard pediatric neurology care

INTERVENTIONS:
Behavioral: Clinic-based and technology-supported sleep intervention — CATS sleep intervention: The in-person sleep education and consultation will consist of 3 face-to-face, one-on-one sessions held 3 months apart during the child's routine clinic visit.The digital component of the sleep intervention will extend in-person education by providing ongoing support. Participants will receive one digital session per week for four weeks after the baseline, 3-month, and 6-month clinic visits, totaling 12 sessions.
  Arms: Experimental intervention group

SUMMARY:
Sleep problems are more common and more severe in children with epilepsy. The purpose of this study is to develop and evaluate the effect of a clinic-based and technology-supported sleep intervention for improving sleep and health in children with epilepsy and their parents.

DETAILED DESCRIPTION:
Participants in the intervention group will receive a standard pediatric neurology care plus a hybrid in-person and digital sleep education program.

ELIGIBILITY:
Inclusion Criteria:

* Children aged between 1.5 and 9 years with a confirmed diagnosis of epilepsy.
* Parents with sufficient Chinese language skills to fully comprehend the trial and complete questionnaires.

Exclusion Criteria:

* Children with cerebral palsy or those who are bedridden.
* Children with a documented sleep disorder, such as obstructive or central sleep apnea and sleep-related movement disorders
* Children born with a congenital, genetic, or orthopedic abnormality that limit their activities of daily living or impair their physical activity.

Ages: 18 Months to 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 150 (Estimated)
Dates: Start 2024-11-19 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Objective sleep parameter by actigraphy | Baseline, 3 , 6 , and 12 months after randomization
  Actigraphy is an objective sleep measurement method that assesses physical motion through a small device worn on the non-dominant wrist. Children's sleep will be objectively assessed for 7 days using actigraphy at each assessment time point. The monitor is a wristwatch-like device with an accelerometer sensitive to body movement. Detected physical motion will be stored as activity counts at 30-second intervals and converted to sleep parameters. Outcome measures derived from actigraphy will include:
  1. sleep quantity variables as measured by durations of nighttime, daytime, and total 24 hour sleep.
  2. sleep quality variable as measured by sleep efficiency.

CONTACTS AND LOCATIONS:
Overall Officials: Shao-Yu Tsai, Principal Investigator — National Taiwan University
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No